CLINICAL TRIAL: NCT06090162
Title: LIBERTY: Liquid Biopsy to Diagnose and Monitor Central Nervous System (CNS) Involvement in High-risk B Cell Non-Hodgkin Lymphoma
Brief Title: LIBERTY: Liquid Biopsy to Diagnose and Monitor CNS Involvement in High-risk B Cell Non-Hodgkin Lymphoma
Acronym: SAKK 38/23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SAKK 38/23
Record Dates: First submitted 2023-10-12; First posted 2023-10-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Non-hodgkin Lymphoma, B Cell
Keywords: High-risk B Cell Non-Hodgkin Lymphoma; ctDNA; experimental diagnostic test
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: This is a multicenter prospective diagnostic study to compare the performance of experimental diagnostic test (ctDNA) versus conventional cytology (CC) and flow cytometry (FC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental diagnostic test (Experimental): Lumbar punction at diagnosis. CSF and blood samples will be assessed by the two diagnostic tests (CSF ctDNA and conventional test (CC/FC))
  Interventions: Diagnostic Test: ctDNA detection

INTERVENTIONS:
Diagnostic Test: ctDNA detection — ctDNA detection on CSF and blood

SUMMARY:
Prevention and treatment of CNS relapse remains a great unmet clinical need in the management of aggressive B-NHL. Hence, investigating novel diagnostic tests is of paramount importance to improve risk-stratification of lymphoma patients at diagnosis, as is the evaluation of novel therapeutic approaches that may prevent and / or treat CNS recurrence. Based on the highlighted evidence, the investigators hypothesize that ctDNA detected within the CSF could potentially improve the detection rate of CNS involvement and consequently improve patients' stratification and better discriminate those in need of consolidative CNS prophylaxis on a molecular basis. Similarly, the investigators postulate that CSF ctDNA could be used as a monitoring tool to assess treatment response and guide therapeutic management.

DETAILED DESCRIPTION:
Non-Hodgkin B-cell lymphoma (B-NHL) are cancers that arise from a subtype of white blood cells (lymphocyte) and typically involve the lymphatic system; they represent 4% of all cancers [SEER database, access 2022]. Despite booming novel antineoplastic agent development, a significant number of aggressive B-NHL patients continue to succumb to their disease, experiencing rapidly progressive disease or early relapse. Central nervous system or CNS (brain, spinal cord and cerebrospinal fluid (CSF)) involvement in aggressive B-NHL is a rare (2-5%) but it is a devastating event, with a life expectancy ranging between 2 and 5 months [PMID: 30125215]. Circulating tumor DNA (ctDNA) represents fragmented DNA that originates from tumors cells, carrying specific cancer-associated mutations that can be detected in the blood or other fluids subsumed under "liquid biopsies".

The role of ctDNA gained momentum with the advent of high throughput sequencing technologies, becoming increasingly relevant for clinical practice. In lymphoma, detecting and monitoring ctDNA has been shown to be feasible and of high prognostic relevance regarding response and relapse. As such, ctDNA is emerging as a promising biomarker that can provide valuable diagnostic and prognostic information [PMID: 30125215, PMID: 29449275]. Identification of patients suffering from aggressive B-NHL at high risk of CNS relapse remains extremely challenging and currently mainly relies on a clinical score (CNS-IPI) [PMID: 27382100]. The detection of asymptomatic CNS is limited to conventional techniques and is not standardized [PMID: 22927246]. In patients with biopsy-proven CNS lymphoma, ctDNA can be detected in CSF (CSF ctDNA) in approximately 95% of cases. Furthermore, CSF ctDNA is predictive of CNS relapse in a small series of neurologically asymptomatic patients with aggressive B-NHL [PMID: 36542815, PMID: 32079701, PMID: 34551072]. Prevention and treatment of CNS involvement remains a great unmet clinical need. The discovery of novel and robust biomarkers is of paramount importance for early detection and risk-adapted therapeutic strategies for CNS involvement. The investigators hypothesize that CSF ctDNA is superior to current standard diagnostic procedures (e.g., flowcytometry or cytology) to detect CNS involvement in high-risk patients.

Furthermore, in patients with positive CSF ctDNA, the investigators also postulate that the concept of monitoring minimal residual disease (MRD, small amount of ctDNA that persists in patients that have no signs of active disease on standard imaging techniques) will provide additional information on patient prognosis.

This is a multicenter prospective diagnostic study to compare the performance of experimental diagnostic test (ctDNA) versus conventional cytology (CC) and flow cytometry (FC). Each high-risk B-NHL participant will proceed through standard work-up to evaluate potential CNS involvement including a neurological physical examination, a brain MRI and a diagnostic lumbar puncture. Each participant's CSF will be assessed by the two diagnostic tests (CSF ctDNA and conventional test (CC/FC)); the gold standard being proven CNS lymphoma involvement.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature before registration and prior to any trial specific procedures, according to Swiss law and ICH E6 regulations Swiss law and ICH GCP E6(R2) regulations before registration.
* Histologically and/or cytologically confirmed newly diagnosed lymphomas including the following:
* Diffuse large B-cell lymphoma (DLBCL) with at least one of the following characteristics:

  * CNS IPI > 4
  * Non-GC/ABC subtype with IPI > 3
  * Testicular involvement
  * Breast involvement
  * Kidney involvement
  * Adrenal involvement
  * Paranasal sinus / orbit involvement
  * Involvement of ≥ 3 extranodal sites
  * HIV-positive
  * Radiological or histological CNS involvement
* High-grade B-cell lymphoma with MYC translocation with BCL2 and / or BCL6 (HGBL)
* Burkitt lymphoma
* Mantle cell lymphoma (blastoid variant or Ki67 >30% or TP53 mutated)
* Primary CNS lymphoma

Note:

* Aggressive transformation from indolent lymphomas (pretreated or not) are allowed
* Patients enrolled in other clinical trials may be included

  * Patients must be willing to undergo a lumbar puncture at screening
  * Age ≥ 18 years

Exclusion Criteria:

* Subtypes of Non-Hodgkin lymphoma (NHL) not fulfilling above mentioned criteria (e.g., indolent lymphoma, T-cell lymphoma)
* Relapsing B-NHL
* Low/intermediate-risk DLBCL (CNS-IPI < 4) AND no CNS involvement on imaging
* Any prior lymphoma-directed therapy before registration, with the exception of a maximum of 48 hours steroids prior to lumbar puncture procedure and therapies received for indolent lymphomas prior to transformation
* Any active advanced or metastatic cancer
* Any clinical contraindication to lumbar puncture procedure as per local guidelines
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned diagnostic procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | at baseline
  Sensitivity of liquid biopsy (ctDNA) measured within CSF in its performance to detect CNS involvement in newly diagnosed high-risk B-NHL in comparison to standard conventional diagnostic approaches (CC / FC). For the evaluation of the primary endpoint, only patients with confirmed CNS involvement at baseline (real positives) will be analyzed. CNS involvement at baseline is defined as having at least one of the following conditions:
  * Positive brain or spine MRI
  * Neurological symptoms of lymphoma manifestations (including ophthalmic symptoms)
  * Histologically confirmed CNS involvement

SECONDARY OUTCOMES:
Specificity | at baseline
  Specificity of liquid biopsy (ctDNA) measured within CSF in its performance to detect CNS involvement in newly diagnosed high-risk B-NHL in comparison to standard conventional diagnostic approaches (CC / FC). For the evaluation of specificity, only patients without CNS involvement at baseline (real negatives) will be analyzed. Absence of CNS involvement at baseline is defined as having none of the following conditions:
  * Positive brain or spine MRI
  * Neurological symptoms of lymphoma manifestations (including ophthalmic symptoms)
  * Histologically confirmed CNS involvement
Time to lymphoma manifestation in the CNS | from the date of registration until the date of assessment of neurological symptoms or death due to lymphoma, assessed up to 1 year after registration
  Time to lymphoma manifestation in the CNS, defined as time from diagnosis to one of the following events, whatever occurs first:
  * Clinical neurological symptoms likely related to lymphoma manifestations
  * Brain or spine MRI changes compatible with lymphoma involvement
  * Histologically confirmed CNS involvement
  * Confirmed involvement of the eye (positive CC / FC)
  * Death due to lymphoma Patients without lymphoma manifestation in the CNS will be censored at their last tumor assessment by CNS imaging showing non-progression
Progression-free survival (PFS) | from the date of registration until the date of progression or relapse as per Lugano and / or IPCG criteria, or death whatever occurs first, assessed up to 1 year after registration
  PFS is defined as the time from diagnosis to lymphoma progression or relapse as per Lugano and / or IPCG criteria, or death whatever occurs first. Patients not having an event at the time of the analysis will be censored at the date of their last tumor assessment showing non-progression.
Event-free survival (EFS) | from the date of registration until the date of progression or relapse as per Lugano and / or IPCG criteria, treatment stop without achieving a complete response or death whatever occurs first, assessed up to 1 year after registration
  EFS is defined as the time from diagnosis to lymphoma progression or relapse as per Lugano and / or IPCG criteria, treatment stop without achieving a complete response or death whatever occurs first. Patients not having an event at the time of analysis will be censored at the date of their last tumor assessment showing non-progression. This endpoint will be calculated separately for each treatment line.
Overall survival (OS) | from the date of registration until the date of death, assessed up to 1 year after registration
  OS will be calculated from diagnosis until death from any cause. Patients not experiencing an event will be censored at the last date they were known to be alive.
Overall response rate (ORR) | At the date of tumor assessment according to the Lugano criteria, assessed up to 1 year after registration
  Overall response rate (ORR) is defined as either PR or CR according to the Lugano criteria. Patients with no tumor assessment will be considered:
  * non-ORR, if they have no following tumor assessment within the trial (patient died, refused or was lost to follow-up) or if they have non-ORR at the following tumor assessment after the end of therapy.
  * ORR, if they have ORR at the following tumor assessment after end of therapy. This endpoint will be calculated separately for each treatment line.
Duration of response (DOR) | from the date of first response CR until the date of lymphoma progression, relapse or death, whatever occurs first, assessed up to 1 years after registration
  DOR is evaluated in all patients who achieved a CR after the end of the intended treatment. DOR is defined as time from first complete response until lymphoma progression, relapse or death, whatever occurs first. Response and progression are evaluated according to Lugano criteria. Patients not having an event at the time of analysis will be censored at the date of their last tumor assessment showing non-progression.
Time to minimal residual disease (MRD) negativity | from the date of first documented MRD positivity (CSF ctDNA detected positive) to the date of first documented MRD negativity, assessed up to 1 years after registration
  Time from first documented MRD positivity (CSF ctDNA detected positive) to first documented MRD negativity. Patients not reaching MRD negativity will be censored at the last time they were known to be MRD positive. Evaluated only in patients with documented MRD positivity at any time.

CONTACTS AND LOCATIONS:
Overall Officials: Noémie Lang, MD, Study Chair — Hôpitaux Universitaires Genève
Locations (14):
- Switzerland (14):
  - Kantonspital Aarau, Aarau
  - Universitätsspital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Inselspital Bern - Universitätsklinik für Medizinische Onkologie, Bern
  - Kantonsspital Graubünden, Chur
  - Hôpital Fribourgeois - Hôpital Cantonal, Fribourg
  - Hopitaux Universitaire de Genève (HUG), Geneva
  - CHUV - Départment d'oncologie, Lausanne
  - Kantonsspital Baselland, Liestal
  - Kantonsspital Münsterlingen, Münsterlingen
  - Kantonsspital St. Gallen, Sankt Gallen
  - Hôpital du Valais, Hôpital de Sion, Sion
  - Klinik für Hämatologie und Onkologie Hirslanden Zürich, Zurich
  - Stadtspital Triemli Zürich, Zurich